CLINICAL TRIAL: NCT00431353
Title: A Randomized, Open-label Study of the Effect of Oral Valcyte Versus Intravenous Ganciclovir on CMV Viremia in Solid Organ Transplant Patients
Brief Title: VICTOR Study - A Study of Valcyte (Valganciclovir po) Compared to Ganciclovir iv in Patients With Cytomegalovirus (CMV) Disease Who Are Solid Organ Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MV17973
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Ganciclovir; Valganciclovir

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: valganciclovir [Valcyte]
- 2 (Experimental)
  Interventions: Drug: Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir — 5mg/kg iv bid for 21 days
  Arms: 2
Drug: valganciclovir [Valcyte] — 900mg po bid for 21 days
  Arms: 1

SUMMARY:
This 2 arm study will evaluate the efficacy and safety of oral Valcyte compared with intravenous ganciclovir for the treatment of CMV disease in solid organ transplant recipients. Eligible patients will be randomized to receive either 1)Valcyte 900mg po bid or 2)ganciclovir 5mg/kg iv bid. The anticipated time on study treatment is 1-2 years and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* recipients of solid organ(s) transplant;
* virologic and clinical evidence of CMV disease after transplantation;
* patients of childbearing potential must be prepared to use effective contraception throughout, and for 90 days after the end of the study.

Exclusion Criteria:

* life-threatening CMV disease according to the investigator's judgment;
* pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2004-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment success (CMV viremia BLQ) | Day 21

SECONDARY OUTCOMES:
Time to eradication of CMV viremia, percentage of patients with resolution of symptoms, percentage of patients with eradication of CMV viremia, time to CMV viremia recurrence, effect on HHV-6, HHV-7 and EBV viremia. | Throughout study
AEs, laboratory parameters, appearance of ganciclovir resistance. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (46):
- Australia (4):
  - Chermside
  - Darlinghurst
  - Sydney
  - Woolloongabba
- Vienna, Austria
- Brussels, Belgium
- Brazil (3):
  - Campinas
  - Porto Alegre
  - São Paulo
- Canada (2):
  - Edmonton, Alberta
  - Toronto, Ontario
- Zagreb, Croatia
- Estonia (2):
  - Tallinn
  - Tartu
- India (4):
  - Chennai
  - Lucknow
  - New Delhi
  - Vellore
- Dublin, Ireland
- Italy (2):
  - Coppito
  - Padua
- Riga, Latvia
- Mexico (2):
  - Aguascalientes
  - Mexico City
- Auckland, New Zealand
- Oslo, Norway
- Poland (6):
  - Bydgoszcz
  - Gdansk
  - Poznan
  - Warsaw
  - Wroclaw
  - Zabrze
- Belgrade, Serbia
- Spain (5):
  - Alicante
  - Barakaldo
  - Barcelona
  - Madrid
  - San Cristóbal de La Laguna
- Basel, Switzerland
- Turkey (Türkiye) (3):
  - Antalya
  - Istanbul
  - Izmir
- United Kingdom (2):
  - Liverpool
  - Oxford
- Venezuela (2):
  - Caracas
  - Maracaibo

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045
- [Derived] Ueland T, Rollag H, Hartmann A, Jardine A, Humar A, Bignamini AA, Asberg A, Aukrust P. Increased osteoprotegerin predicts poor virological outcome during anticytomegalovirus therapy in solid organ transplant recipients. Transplantation. 2015 Jan;99(1):100-5. doi: 10.1097/TP.0000000000000227. PMID 24983306
- [Derived] Ueland T, Rollag H, Hartmann A, Jardine AG, Humar A, Michelsen AE, Bignamini AA, Asberg A, Aukrust P. Secreted Wnt antagonists during eradication of cytomegalovirus infection in solid organ transplant recipients. Am J Transplant. 2014 Jan;14(1):210-5. doi: 10.1111/ajt.12506. Epub 2013 Nov 13. PMID 24224707
- [Derived] Rollag H, Ueland T, Asberg A, Hartmann A, Jardine AG, Humar A, Pescovitz MD, Bignamini AA, Aukrust P. Characterization of cytomegalovirus disease in solid organ transplant recipients by markers of inflammation in plasma. PLoS One. 2013 Apr 8;8(4):e60767. doi: 10.1371/journal.pone.0060767. Print 2013. PMID 23593305
- [Derived] Razonable RR, Asberg A, Rollag H, Duncan J, Boisvert D, Yao JD, Caliendo AM, Humar A, Do TD. Virologic suppression measured by a cytomegalovirus (CMV) DNA test calibrated to the World Health Organization international standard is predictive of CMV disease resolution in transplant recipients. Clin Infect Dis. 2013 Jun;56(11):1546-53. doi: 10.1093/cid/cit096. Epub 2013 Feb 15. PMID 23418272